CLINICAL TRIAL: NCT02780427
Title: ED50 and ED95 of Intranasal Dexmedetomidine in Pediatric Patients Undergoing Transthoracic Echocardiography Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Wenhua Zhang, Director, Clinical Resesearch, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Wzhang03
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Patients for Transthoracic Echocardiography; Unknown Diagnosis
Keywords: Dose-Response Relationship, Drug

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1-6 months (Group 1) (Active Comparator)
  Interventions: Drug: intranasal dexmedetomidine
- 7-12 months (Group 2) (Active Comparator)
  Interventions: Drug: intranasal dexmedetomidine
- 13-18 months (Group 3) (Active Comparator)
  Interventions: Drug: intranasal dexmedetomidine
- 19-24 months (Group 4) (Active Comparator)
  Interventions: Drug: intranasal dexmedetomidine

INTERVENTIONS:
Drug: intranasal dexmedetomidine — Phase 1, Children received a bolus of intranasal dexmedetomidine which adjusted by the "Dixon up-and-down method for TEE study. The first child received 2.5 mcg/kg of intranasal dexmedetomidine dose (100mcg/ml), and the dose varied by 0.1 mcg/kg according to the up-and-down method Phase 2 was a dose-escalation study. After interim analysis of the phase 1 results, four dose levels above the calculated ED50 were defined. Dose spacing was set at 0.25 mcg/kg of intranasal dexmedetomidine consistent with the re-estimated standard deviation (SD).

SUMMARY:
The median effective dose (ED50) and ED95 of intranasal dexmedetomidine as a single bolus have not been described for sedation in children undergoing transthoracic echocardiography (TEE) study. This information is important to compare agents and to determine the most effective sedative dose. The investigators performed a two-stage study to determine the ED50 and the ED95 of intranasal dexmedetomidine to investigate age-related differences in participants undergoing transthoracic echocardiography study.

DETAILED DESCRIPTION:
The investigators performed a two-stage study to determine the ED50 and the ED95 of intranasal dexmedetomidine in children undergoing transthoracic echocardiography study. In phase 1, 120 participants were randomized in a Dixon-Massey study to describe the minimum local sedative dose. In phase 2, a further 160 participants were randomly allocated to receive sedation with doses in the upper dose-response range to define the ED95

ELIGIBILITY:
Inclusion Criteria:

* Children, aged between one and 24 months. classified as (American Society of Anesthesiologists) ASA physical status I or II, undergoing TEE were enrolled in the study.

Exclusion Criteria:

* Known allergy or hypersensitive reaction to dexmedetomidine
* Organ dysfunction, and significant developmental delays or behavior problems
* Cardiac arrhythmia
* Known. acyanotic congenital heart disease or children after cardiac interventional procedures for follow-up examination.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
The ED50 doses for intranasal dexmedetomidine | up to 0.5 hours after transthoracic echocardiography
  Phase 1: The starting dose of dexmedetomidine was 2.5 mcg/kg. These doses varied by 0.1 mcg/kg, according to the up-and-down method 18. If the detected MOAA/S score was >3 within 45 minutes after intranasal administration, or clinically adequate diagnostic-quality images could not be acquired, sedation was considered a failure; and the dexmedetomidine dose was increased by 0.1 mcg/kg in the next patient of the same age group. In contrast, if the detected MOAA/S score was ≤3 and the acquisition of clinically adequate diagnostic-quality images was possible, the sedation was considered successful; and the dexmedetomidine dose was decreased by 0.1 mcg/kg in the next patient o
The ED95 doses for intranasal dexmedetomidine | up to 0.5 hours after transthoracic echocardiography
  Phase 2 was a dose-escalation study. After interim analysis of the phase 1 results, four dose levels above the calculated ED50 were defined. Dose spacing was set at 0.3 mcg/kg of intranasal dexmedetomidine consistent with the re-estimated standard deviation (SD). Defined levels were set at about 2.5, 2.75, 3.0, and 3.25 mcg/kg of intranasal dexmedetomidine. Criteria for success and failure were identical to those in phase 1.
  Successful sedation was defined as a MOAA/S score between 0-3 and allowed the acquisition of clinically adequate diagnostic-quality images, while failure was defined as a MOAA/S score >3 within 45 minutes or clinically adequate diagnostic-quality images could not be acquired
Score of physical movement | up to 0.5 hours after transthoracic echocardiography
  Movement score was recorded by sonographers who were blinded to the sedative regimen.
  1. No movement
  2. Occasional, slight movement
  3. Frequent, slight movement
  4. Vigorous movement limited to extremities
  5. Vigorous movement, including torso and head

SECONDARY OUTCOMES:
sedation induction time | up to 2 hours after drug administration
  Successful sedation was defined as an MOAA/S of between 0 and 3, and sedation induction time was defined as the time from drug administration to the onset of satisfactory sedation
Wake -up time | up to 2 hours after drug administration
  Children were classified as awake if the MOAA/S was between 4 and 6. Wake -up time was defined as the time from successful sedation until the time that the child awoke

OTHER OUTCOMES:
heart rate | up to 3 hours after drug administration
  Bradycardia was defined as a reduction in heart rate more than 20% from the baseline values
Oxyhemoglobin desaturation | up to 3 hours after drug administration
  Significant Oxyhemoglobin desaturation was defined as < 90%.
non-invasive systolic blood pressure | up to 3 hours after drug administration
  Hypotension was defined as a reduction in systolic blood pressure more than 20% from the baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology of Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China